CLINICAL TRIAL: NCT03210896
Title: Breath for Better Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RA315217
Record Dates: First submitted 2017-06-21; First posted 2017-07-07 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Main Group (No Intervention): 100 subjects (70 T2D and 30 Controls) consent to provide 1 venous blood sample, 1 capillary blood sample and 3 breath samples using IMSPEX, Bio-VOC and ReCIVA breath samplers.
- Sub Group I (Experimental): 20 subjects from the main group (10 T2D and 10 Controls) to remain after providing the above samples. These patients will stay for an additional 3 hours and provide 1 capillary blood sample and 3 breath samples using IMSPEX, Bio-VOC and ReCIVA breath samplers at the following time intervals: 5, 30, 60, 120 & 180 minutes.
  Interventions: Dietary Supplement: Orange juice
- Sub Group II (No Intervention): 5 control subjects consent to provide 1 venous blood sample, 1 capillary blood sample and 3 breath samples using IMSPEX, Bio-VOC and ReCIVA breath samplers. This will be followed by 1 capillary blood sample and 3 breath samples every hour for a total of 5 hours.

INTERVENTIONS:
Dietary Supplement: Orange juice — Sub group I will drink Orange juice and have repeat measures.
  Arms: Sub Group I

SUMMARY:
Breath analysis is becoming of increasing interest to researchers throughout the world for disease identification and monitoring. It is known that small chemicals dissolved in the blood can pass through the blood/air barrier within the lungs and be exhaled in normal breath, with many of these chemicals being potential biomarkers for a broad range of diseases. These specific biomarkers need to be identified so that gas analysis instruments and sensors can be designed to detect these chemicals.

The aim of this study is to determine if there are biomarkers in exhaled breath that correlate with blood glucose concentration. This biomarker can then be used to produce a new device that will allow diabetic patients to monitor their blood glucose levels in a quick and non-invasive way. The investigators believe this will lead to a significant improvement in the quality of life of those suffering from this condition.

In this study breath samples will be collected using three different methods to maximise the chemical information available from each breath. Breath samples from Type 2 diabetic patients will be compared with healthy controls. Subgroups will have repeated breath samples after drinking orange juice or during normal day-to-day activities. This is to measure any changes in breath chemicals over time. The chemicals detected will be compared with blood tests, to identify potential breath biomarkers for blood glucose concentration, and to see if factors such as sex, age, and diet have any effect on the biomarkers detected.

This is a single centre pilot study taking place at University Hospitals Coventry and Warwickshire NHS Trust, and the analysis of the breath samples will be carried out at the University of Warwick.

DETAILED DESCRIPTION:
Breath analysis is becoming of increasing interest to researchers throughout the world for disease identification and monitoring. It is known that small chemicals dissolved in the blood can pass through the blood/air barrier within the lungs and be exhaled in normal breath, with many of these chemicals being potential biomarkers for a broad range of diseases.

As a biological waste media, it has many advantages over other more invasive approaches. It can be given at will with a large volume of potential sample, it has a high level of patient acceptability, it is non-invasive, sample collection is very quick and it is potentially possible to analyse the sample in almost real-time. This has made breath analysis a target focus for many groups working on a broad range of diseases. Previous studies, by the investigators group and others have shown that breath analysis can be used to identify patients with irritable bowel diseases, hepatic encephalopathy, cancers (specifically colorectal and breast) and respiratory infections (such as tuberculosis).

Though these previous projects have shown promise, it is only now that our ability to make highly sensitive gas analysis instruments and sensors makes it a real possibility to bring this to the wider public. However, to be able to develop such sensors and sensor systems, the investigators need to identify the specific chemical biomarkers in the breath to detect and measure. At this point in time, there is no such definitive list of biomarkers (potential or otherwise) for all possible disease groups. In addition, where there are proposed markers, there is no agreement in the field on what these are.

The final goal of this project is to produce a new device that will allow simple, non-invasive monitoring of diabetic patients, which the investigators believe will lead to a significant improvement in the quality of life of those suffering from this condition.

The purpose of this study is partly to discover new potential biomarkers in human breath associated with diabetes and from this, try and understand what confounding factors may affect its efficacy. The investigators believe that these confounding factors maybe sex, age, diet and food and others. Without a deep understanding of these variables, it will be impossible to develop a new generation of person monitoring tools.

To maximise the chances of discovering new potential biomarkers, the investigators will deploy a range of different analytical instruments aimed at different parts of the chemical spectrum. Together, the investigators believe they will be able to get a comprehensive understanding of the chemicals being released in human breath, how these are affected by confounding factors and how they are related to blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed clinically with type 2 diabetes

Exclusion Criteria:

* Consumed alcohol less than 48 hours before the start of the study appointment
* Consumed food or drink less than 1 hour before the start of the study appointment
* Smoked less than 2 hours before the start of the study appointment
* Pregnant
* Person who has (or had in the last week) a respiratory infection (either bacterial or viral)
* Uses recreational drugs
* Those who have had surgery/major injury in the last 4 months
* Anyone with a different metabolic, liver, cancer or gastro related disease
* Anyone who is taking part in an interventional study
* Anyone who is unable to provide written consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
Chemical components in breath samples will be measured using Ion Mobility Spectrometry, to determine if there are potential biomarkers in exhaled breath that can be directly correlated with blood glucose concentration. | Baseline, 5 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours.
  Repeat breath samples will be collected over time to measure changes in chemical components.
Chemical components in breath will be captured into a plastic tubes (Bio-VOC) followed by Electronic Nose analysis, to determine if there are potential biomarkers in exhaled breath that can be directly correlated with blood glucose concentration. | Baseline, 5 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours.
  Repeat breath samples will be collected over time to measure changes in chemical components.
Chemical components in breath will be captured into absorbent tubes followed by GCMS analysis, to determine if there are potential biomarkers in exhaled breath that can be directly correlated with blood glucose concentration. | Baseline, 5 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours.
  Repeat breath samples will be collected over time to measure changes in chemical components.

SECONDARY OUTCOMES:
Demographic and lifestyle data will be recorded to see if they correlate with breath chemical composition. | Baseline
  Confounding factors such as age will be recorded to see if they influence the breath chemical composition.
Demographic and lifestyle data will be recorded to see if they correlate with breath chemical composition. | Baseline
  Confounding factors such as sex will be recorded to see if they influence the breath chemical composition.
Demographic and lifestyle data will be recorded to see if they correlate with breath chemical composition. | Baseline
  Confounding factors such as smoking habits will be recorded to see if they influence the breath chemical composition.
Demographic and lifestyle data will be recorded to see if they correlate with breath chemical composition. | Baseline
  Confounding factors such as medication will be recorded to see if they influence the breath chemical composition.
Demographic and lifestyle data will be recorded to see if they correlate with breath chemical composition. | Baseline
  Confounding factors such as food intake will be recorded to see if they influence the breath chemical composition.
Demographic and lifestyle data will be recorded to see if they correlate with breath chemical composition. | Baseline
  Confounding factors such as physical activities will be recorded to see if they influence the breath chemical composition.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Arasaradanam, Principal Investigator — Consultant
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arasaradnam RP, McFarlane M, Daulton E, Skinner J, O'Connell N, Wurie S, Chambers S, Nwokolo C, Bardhan K, Savage R, Covington J. Non-invasive exhaled volatile organic biomarker analysis to detect inflammatory bowel disease (IBD). Dig Liver Dis. 2016 Feb;48(2):148-53. doi: 10.1016/j.dld.2015.10.013. Epub 2015 Nov 22. PMID 26682719
- [Background] Arasaradnam RP, McFarlane M, Ling K, Wurie S, O'Connell N, Nwokolo CU, Bardhan KD, Skinner J, Savage RS, Covington JA. Breathomics--exhaled volatile organic compound analysis to detect hepatic encephalopathy: a pilot study. J Breath Res. 2016 Feb 11;10(1):016012. doi: 10.1088/1752-7155/10/1/016012. PMID 26866470
- [Background] Amal H, Leja M, Funka K, Lasina I, Skapars R, Sivins A, Ancans G, Kikuste I, Vanags A, Tolmanis I, Kirsners A, Kupcinskas L, Haick H. Breath testing as potential colorectal cancer screening tool. Int J Cancer. 2016 Jan 1;138(1):229-36. doi: 10.1002/ijc.29701. Epub 2015 Aug 7. PMID 26212114
- [Background] Phillips M, Cataneo RN, Ditkoff BA, Fisher P, Greenberg J, Gunawardena R, Kwon CS, Tietje O, Wong C. Prediction of breast cancer using volatile biomarkers in the breath. Breast Cancer Res Treat. 2006 Sep;99(1):19-21. doi: 10.1007/s10549-006-9176-1. Epub 2006 Feb 24. PMID 16502014
- [Background] Sahota AS, Gowda R, Arasaradnam RP, Daulton E, Savage RS, Skinner JR, Adams E, Ward SA, Covington JA. A simple breath test for tuberculosis using ion mobility: A pilot study. Tuberculosis (Edinb). 2016 Jul;99:143-146. doi: 10.1016/j.tube.2016.05.005. Epub 2016 May 29. PMID 27450016